CLINICAL TRIAL: NCT03481855
Title: Plethysmographic Pulse-contour and Pulse-wave-transit-times for Haemodynamic Evaluation in Bleeding Simulation
Acronym: Plethysmo
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Technische Universität Berlin (Other)
Responsible Party: Principal Investigator, Aarne Feldheiser, Priv.-Doz. Dr. med. Aarne Feldheiser, Charite University, Berlin, Germany
Other Study IDs: EA1/249/17
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Health, Subjective

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Progressive bleeding simulation: The study intervention by a lower-body-low-pressure chamber is performed in this group of healthy volunteers with progressive increase of negative pressure by a step-wise approach (-15mmHg, -30mmHg, -45mmHg).
  Interventions: Device: Lower-body-low-pressure chamber
- Prolonged bleeding simulation: The study intervention by a lower-body-low-pressure chamber is performed in this group of healthy volunteers with prolonged exposure to a negative pressure of -15mmHg.
  Interventions: Device: Lower-body-low-pressure chamber

INTERVENTIONS:
Device: Lower-body-low-pressure chamber — The lower-body-low-pressure chamber administers a negative pressure to the lower part of the body (below the waist) to induce a central hypovolaemia by pooling of blood in the legs according to Tymko, M. FACETS, Bd. 1, Nr. 1, S. 225-244, März 2017 and Esch, B.T.A. et al. AJP Adv. Physiol. Educ., Bd. 31, Nr. 1, S. 76-81, März 2007.

SUMMARY:
The evaluation of haemodynamic changes is still challenging in clinically relevant situations (e.g. in bleeding, septic and postoperative patients) with the conventional monitoring routinely used including heart rate and mean arterial pressure. If the arterial pressure drops and the heart increases, the haemodynamic state is already decompensated and a therapy is at risk being indicated too late.

Prior to decompensation - still in the state of compensated shock - it would be desirable to detect the shock already. The compensated shock is characterized by an occult drop of cardiac output and a hypoperfusion of vital organs like e.g. the splanchnic region. Due to these pathophysiological characteristics, a therapy would be indicated already in this stadium of shock progression.

The available monitoring tools to detect compensated shock are on the one hand side invasive (intravascular catheter), cost-intensive (cost of the catheter systems), or need extensive training (echocardiography). Consequently, the implementation of advanced haemodynamic monitoring is still low despite the high clinical relevance for the patients.

It is the goal of this project to evaluate in healthy volunteers the routinely implemented technology of photo-plethysmography in its ability to detect haemodynamic changes by extended signal analysis of the pulse-contour and the pulse-wave-transit-times in relation to the gold-standard echocardiography.

Secondary goal of this study is to analyse the physiological and haemodynamic changes during progressive central hypovolaemia displayed by non-invasive or minimal-invasive monitoring devices and associate the changes to each other.

ELIGIBILITY:
Inclusion Criteria:

* Offered patient information and written informed consent
* Existence of valid health insurance
* Male gender

Exclusion Criteria:

* Patients aged less than 18 years or more than 40 years
* Inability of German language use
* Lacking willingness to save and hand out data within the study
* Evidence of a chronic disease (cardio-vascular, renal, pulmonary, neurological, metabolic, gastro-intestinal)
* Chronic medication
* Signs of a reduced cardiorespiratory capacity
* Signs of an acute illness
* Participation in a prospective intervention trial during the study period
* Anamnestic hints for syncope or disposition to hypotension
* Signs of arterial hypertension
* Signs of inguinal hernia
* Relevant pathologies in the baseline examination of the transthoracic echocardiography
* For the bio-impedance measurements: heart defibrillator

Ages: 18 Years to 40 Years | Sex: Male
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Changes in the pulse-contour-analysis of the plethysmographic signal | Time course of 40 minutes (at study baseline, at study intervention level 1, 2 and 3 and recovery time)
  The pulse-contour of the plethysmographic signal will be analyzed to detect morphological changes over time in relation to the initial baseline recording
Changes the pulse-wave-transit-times of the plethysmographic signal | Time course of 40 minutes (at study baseline, at study intervention level 1, 2 and 3 and recovery time)
  The pulse-wave-transit-times of the plethysmographic signal will be analyzed to detect changes over time in relation to the initial baseline recording

SECONDARY OUTCOMES:
Arterial blood pressure | At baseline (up to minute 7 after starting the study protocol), during the study intervention level 1, 2 and 3 (between minute 8 up to minute 28 after starting study protocol) and recovery after finishing the study intervention (between minute 30 and 40)
  Arterial blood pressure determined by non-invasive monitoring
Heart rate | At baseline (up to minute 7 after starting the study protocol), during the study intervention level 1, 2 and 3 (between minute 8 up to minute 28 after starting study protocol) and recovery after finishing the study intervention (between minute 30 and 40)
  Heart rate determined by non-invasive monitoring
Echocardiographic parameter to determine the cardiac performance of the left ventricle | At baseline (up to minute 7 after starting the study protocol), during the study intervention level 1, 2 and 3 (between minute 8 up to minute 28 after starting study protocol) and recovery after finishing the study intervention (between minute 30 and 40)
  The performance of the left ventricle will be analyzed by a transthoracic echocardiography by a physician certified by the European Society of Cardiology
Echocardiographic parameter to determine the cardiac performance of the left atrium | At baseline (up to minute 7 after starting the study protocol), during the study intervention level 1, 2 and 3 (between minute 8 up to minute 28 after starting study protocol) and recovery after finishing the study intervention (between minute 30 and 40)
  The performance of the left atrium will be analyzed by a transthoracic echocardiography by a physician certified by the European Society of Cardiology
Echocardiographic parameter to determine the cardiac performance of the right ventricle | At baseline (up to minute 7 after starting the study protocol), during the study intervention level 1, 2 and 3 (between minute 8 up to minute 28 after starting study protocol) and recovery after finishing the study intervention (between minute 30 and 40)
  The performance of the right ventricle will be analyzed by a transthoracic echocardiography by a physician certified by the European Society of Cardiology
Echocardiographic parameter to determine the cardiac performance of the right atrium | At baseline (up to minute 7 after starting the study protocol), during the study intervention level 1, 2 and 3 (between minute 8 up to minute 28 after starting study protocol) and recovery after finishing the study intervention (between minute 30 and 40)
  The performance of the right atrium will be analyzed by a transthoracic echocardiography by a physician certified by the European Society of Cardiology
Echocardiographic parameter to analyze the vena cava inferior | At baseline (up to minute 7 after starting the study protocol), during the study intervention level 1, 2 and 3 (between minute 8 up to minute 28 after starting study protocol) and recovery after finishing the study intervention (between minute 30 and 40)
  The analysis will be assessed by a subcostal approach by transthoracic echocardiography
Heart rate variability | At baseline (up to minute 7 after starting the study protocol), during the study intervention level 1, 2 and 3 (between minute 8 up to minute 28 after starting study protocol) and recovery after finishing the study intervention (between minute 30 and 40)
  Heart rate variability calculated from raw biosignals Bioelectrical signals by standardized analysis algorithms
Haemodynamic parameter of the bio-impedance monitoring | Time course of 40 minutes (at study baseline, at study intervention level 1, 2 and 3 and recovery time)
  The parameter will be determined by the electrical cardiometry/bio-impedance monitoring device of Osypka Medical
Shock indices of the bio-impedance monitoring | Time course of 40 minutes (at study baseline, at study intervention level 1, 2 and 3 and recovery time)
  The parameter will be determined by the electrical cardiometry/bio-impedance monitoring device of Osypka Medical
Heart sounds | Time course of 40 minutes (at study baseline, at study intervention level 1, 2 and 3 and recovery time)
  Heart sounds measured by vibration sensors
Tonometric arterial blood pressure | Time course of 40 minutes (at study baseline, at study intervention level 1, 2 and 3 and recovery time)
  Tonometric arterial blood pressure measured by applanation tonometer
Haemodynamic parameter of the tonometric pulse-contour method | Time course of 40 minutes (at study baseline, at study intervention level 1, 2 and 3 and recovery time)
  The parameter will be determined by the non-invasive monitoring device Finapress
Mean systemic filling pressure | At baseline (up to minute 7 after starting the study protocol), during the study intervention level 1, 2 and 3 (between minute 8 up to minute 28 after starting study protocol) and recovery after finishing the study intervention (between minute 30 and 40)
  The parameters describing the characteristics of the venous return determined by the stop-flow method
Questionnaire regarding alimentation | Immediately prior to the start of the study protocol
  The questionnaire directs to characterize the intake of fluid and solid alimentation prior to the study protocol
Bio-impedance analysis of the body fluid | Immediately prior to the start of the study protocol
  The bio-impedance analysis of the body fluid directs to determine the water content of the body

CONTACTS AND LOCATIONS:
Overall Officials: Aarne Feldheiser, MD, PhD, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Campus Charité Mitte and Campus Virchow Klinikum, Charité - University Medicine Berlin Berlin, Germany, 13353 Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Charité Mitte and Campus Virchow Klinikum, Charité - University Medicine Berlin Berlin, Germany, Berlin, Germany

REFERENCES:
- [Derived] Feldheiser A, Juhl-Olsen P, Nordine M, Stetzuhn M, Wiegank L, Knebel F, Treskatsch S, Berger C. A comprehensive echocardiographic analysis during simulated hypovolaemia: An observational study. Eur J Anaesthesiol. 2023 Aug 1;40(8):578-586. doi: 10.1097/EJA.0000000000001863. Epub 2023 Jun 1. PMID 37265333